CLINICAL TRIAL: NCT02316587
Title: Assessment of Myocardial Fibrosis - Impact on Postoperative Outcome i Patients With Severe Aortic STenosis Undergoing Aortic Valve Replacement
Brief Title: Assessment of Myocardial Fibrosis in Aortic STenosis
Acronym: AMFAST
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Carter-Storch, MD, Odense University Hospital
Other Study IDs: AMFAST
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Endomyocardial Fibrosis; Aortic Valve Stenosis
Keywords: Computerized Tomography; Magnetic Resonance Imaging; Echocardiography; Right Heart Catheterization
MeSH Terms: conditions — Endomyocardial Fibrosis; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma saved for biomarkers Endomyocardial biopsy Stenotic aortic valve
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational cohort study studies the impact myocardial fibrosis has on patients with severe aortic stenosis undergoing aortic valve replacement.

DETAILED DESCRIPTION:
Aortic stenosis is the most common valvular disease in the Western World. It is a slow evolving degenerative disease caused by gradual accumulation of calcium in the valve. Untreated it is fatal. Reduced opening area of the valve increases afterload on the left ventricle (LV), which leads to raised end-diastolic pressure in the LV. Increased wall stress leads to LV hypertrophy and expansion of the extracellular matrix. An abnormally high extracellular volume fraction is called myocardial fibrosis (MF), which causes increased LV stiffness, diastolic dysfunction, dilatation of the left atrium and in the end heart failure.

The standard of treatment for aortic stenosis is an operation, aortic valve repair (AVR), where a mechanical or biological valve replaces the old one. The operation involves a substantial risk of postoperative mortality, and is therefore delayed until the patient develops symptoms such as shortness of breath, chest pains or syncope. For most patients AVR causes significant symptom reduction and reduced mortality. Recent studies have indicated that patient with severe MF, which may account for up to one third of the patients treated, have little or no symptom improvement and an increased mortality after AVR. This raises concern that their LV is so severely fibrotic that it is beyond repair. These patients may not benefit from an operation, or should possibly have had AVR performed at an earlier stage of the disease.

Today, cardiac fibrosis can be detected by a biopsy which is invasive. Late Gadolinium and T1-mapping cardiac Magnetic Resonance imaging (MRi) has recently been evaluated as a new method to detect MF, but this method is costly and contraindicated for some patients. Cardiac Computerized Tomography (CT) has been proposed as a method to evaluate MF, but has not been properly validated yet.

In this study we compare different methods (biopsy, MRi, CT, echocardiography and different biomarkers) to evaluate the extent of MF in 130 patients with severe aortic stenosis undergoing AVR. We will focus on their symptom improvement and survival rate one year after the operation. Our main thesis is that patients with severe fibrosis before the operation have little or no symptom improvement and reduced survival after the operation. If this thesis is correct, it will question which patients to offer AVR. Some patients we operate today may have no benefit from the operation because the left ventricle is damaged from severe fibrosis, and some patients from who we withhold the operation today because they are asymptomatic may benefit from AVR before they develop severe fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic valve stenosis (AVA ≤1cm2).
* Scheduled for aortic valve replacement.
* Signed consent

Exclusion Criteria:

* At least moderate mitral regurgitation or stenosis.
* Primary aortic insufficiency.
* Persistent or permanent atrial fibrillation/flutter.
* CKD with e-GFR < 40 ml/kg/min.
* Pacemaker or Implantable Cardioverter Defibrillator (ICD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe aortic valve stenosis.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
MACE (Major Adverse Cardiac Event) | 2 years
  Major Adverse Cardiac Event defined as all-cause mortality or admission with heart failure

SECONDARY OUTCOMES:
Cardiovascular mortality | 2 years

OTHER OUTCOMES:
NYHA change | 1 year
  New York Heart Association classification of dyspnea
Functional capacity assessed by right heart catheterization and VO2-max test | 1 year
  Functional capacity assessed by right heart catheterization and VO2-max test
Extracellular volume quantification Assessed by biopsy, CT and MRi | 1 year
  Assessed by biopsy, CT and MRi at baseline and after one year
Duke Activity Score Index | 1 year
  Duke Activity Score Index Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Jacob E Møller, MD PhD DMsc, Study Director — Odense University Hospital; Jordi S Dahl, MD, Ph.D., Study Chair — Odense University Hospital; Kristian A Øvrehus, MD, Ph.D., Study Chair — Odense University Hospital; Lars M Rasmussen, MD PhD DMsc, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Derived] Carter-Storch R, Mortensen NSB, Christensen NL, Ali M, Laursen KB, Pellikka PA, Moller JE, Dahl JS. First-phase ejection fraction: association with remodelling and outcome in aortic valve stenosis. Open Heart. 2021 Feb;8(1):e001543. doi: 10.1136/openhrt-2020-001543. PMID 33574022
- [Derived] Carter-Storch R, Dahl JS, Christensen NL, Pecini R, Sondergard EV, Ovrehus KA, Moller JE. Postoperative atrial fibrillation after aortic valve replacement is a risk factor for long-term atrial fibrillation. Interact Cardiovasc Thorac Surg. 2019 Sep 1;29(3):378-385. doi: 10.1093/icvts/ivz094. PMID 30977792
- [Derived] Carter-Storch R, Moller JE, Christensen NL, Irmukhadenov A, Rasmussen LM, Pecini R, Ovrehus KA, Sondergard EV, Marcussen N, Dahl JS. Postoperative Reverse Remodeling and Symptomatic Improvement in Normal-Flow Low-Gradient Aortic Stenosis After Aortic Valve Replacement. Circ Cardiovasc Imaging. 2017 Dec;10(12):e006580. doi: 10.1161/CIRCIMAGING.117.006580. PMID 29222121